CLINICAL TRIAL: NCT04506788
Title: Assessment of EEG Slow Wave Activity in Comatose Cardiac Arrest Survivors Under Propofol Anesthesia
Brief Title: EEG Slow Wave Activity in Hypoxic Brain Injury
Acronym: BrainICU
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Cerenion Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 68/2012
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Cardiac Arrest
Keywords: EEG; Intensive Care; Propofol
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BrainICU is a prospective observational study investigating the EEG slow wave activity in comatose cardiac arrest survivors under propofol anesthesia and its association with neurological outcome.

DETAILED DESCRIPTION:
BrainICU is a prospective observational study investigating the EEG slow wave activity in comatose cardiac arrest survivors under propofol anesthesia and its association with neurological outcome. Comatose adult patients admitted to intensive care unit (ICU) after cardiac arrest are included. Patients with previous neurological disease expected to affect substantially the EEG are excluded. The patients' relatives are asked for an informed written consent to participate. In the intensive care, the patients are sedated using continuous infusion of propofol while receiving temperature management/hypothermia treatment following the ICUs' common practice. EEG is recorded within the first 24h after ICU admission. If possible, the recording is repeated on the second and third day i.e. 48h and 72h after ICU admission, respectively. To induce the maximum effect of propofol on EEG, additional boluses of propofol during the EEG recording may be given until the burst suppression level is reached. Slow wave activity is calculated offline from the EEG recordings. The neurological recovery of the patients is defined 6 months after cardiac arrest from patient documents and/or by phone call to the patient/ relative using Cerebral Performance Category. After the follow-up period patient or the relative is also asked to fill a survey (SF-36) to estimate the health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Comatose patients admitted to intensive care after cardiac arrest

Exclusion Criteria:

* Previous neurological disease expected to affect EEG substantially

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients admitted to intensive care in the study units.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
EEG slow wave activity | 0-72 hours
  EEG slow-wave activity determined from the low-frequency (<1 Hz) signal component calculated from the EEG recordings made within 24 hours from ICU admission and repeated, if possible, at 48 hours and 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kortelainen, MD, PhD, Principal Investigator — University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kortelainen J, Vayrynen E, Juuso I, Laurila J, Koskenkari J, Ala-Kokko T. Forehead electrodes sufficiently detect propofol-induced slow waves for the assessment of brain function after cardiac arrest. J Clin Monit Comput. 2020 Feb;34(1):105-110. doi: 10.1007/s10877-019-00282-3. Epub 2019 Feb 20. PMID 30788811
- [Background] Kortelainen J, Vayrynen E, Huuskonen U, Laurila J, Koskenkari J, Backman JT, Alahuhta S, Seppanen T, Ala-Kokko T. Pilot Study of Propofol-induced Slow Waves as a Pharmacologic Test for Brain Dysfunction after Brain Injury. Anesthesiology. 2017 Jan;126(1):94-103. doi: 10.1097/ALN.0000000000001385. PMID 27749312